CLINICAL TRIAL: NCT04319237
Title: Axicabtagene Ciloleucel:Neurocognitive and Patient-Reported Outcomes
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Other Study IDs: MCC-20372
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B Cell Lymphoma; Transformed Lymphoma
Keywords: Axi-cel therapy; CAR-T
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Neuropsychological Tests; Surveys and Questionnaires; Quality of Life; Costs and Cost Analysis; Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants
  Interventions: Other: Handgrip strength test; Behavioral: Neuropsychological Assessment - Wechsler Test of Adult Reading (WTAR); Behavioral: Neuropsychological Assessment - Repeatable Battery for the Assessment of Status (RBANS); Behavioral: Neuropsychological Assessment - Color Trails; Behavioral: Neuropsychological Assessment -Stroop Color and Word Test; Behavioral: Patient Reported Outcomes Measurement Information System-29 (PROMIS-29) Questionnaire; Behavioral: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire; Behavioral: Quality of Life (EQ-5D-5L) Questionnaire; Behavioral: PROMIS Cognitive Function 4a Questionnaire; Behavioral: Comprehensive Score for Financial Toxicity (COST) measure

INTERVENTIONS:
Other: Handgrip strength test — The purpose of this test is to measure the maximum isometric strength of the hand and forearm muscles.
Behavioral: Neuropsychological Assessment - Wechsler Test of Adult Reading (WTAR) — The Wechsler Test of Adult Reading (WTAR) is a neuropsychological assessment tool used to provide a measure of Intellectual function. Participants are presented with 50 irregularly spelled words and prompted to pronounce each; the irregular grapheme-to-phoneme translations (such as the "gh" in the word tough) in the prompts make it difficult to pronounce without having previously learned the word. A high WTAR score is correlated with higher general intelligence as measured by the Wechsler intelligence scales.
Behavioral: Neuropsychological Assessment - Repeatable Battery for the Assessment of Status (RBANS) — The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) consists of twelve subtests which give five scores, one for each of the five domains tested (immediate memory, visuospatial/constructional, language, attention, delayed memory).
Behavioral: Neuropsychological Assessment - Color Trails — The Color Trails test measures sustained attention and sequencing. Numbered circles are printed with vivid pink or yellow backgrounds that are perceptible to color-blind individuals. Participants rapidly connect circles numbered 1-25 in sequence and rapidly connect numbered circles in sequence, but alternates between pink and yellow. The length of time to complete each trial is recorded, along with qualitative features of performance indicative of brain dysfunction, such as near-misses, prompts, number sequence errors, and color sequence errors.
Behavioral: Neuropsychological Assessment -Stroop Color and Word Test — The Stroop Color and Word Test is based on the observation that individuals can read words much faster than they can identify and name colors. The test-taker reads color words or names ink colors from different pages as quickly as possible within a time limit. The test yields three scores based on the number of items completed on each of the three stimulus sheets. An Interference score is useful in determining the individual's cognitive flexibility, creativity, and reaction to cognitive pressures.
Behavioral: Patient Reported Outcomes Measurement Information System-29 (PROMIS-29) Questionnaire — The PROMIS-29 questionnaire assesses each of 7 domains (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities). A higher score equals more of the concept being measured.
Behavioral: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire — European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C-3) and the add-on EORTC QLQ Non-Hodgkin's Lymphoma (EORTC QLQ-NHL-HG29) module. All scales range from 0-100, a high scale score represents a higher response level. For example, a high functional score represents a high level of functioning.
Behavioral: Quality of Life (EQ-5D-5L) Questionnaire — The EQ-5D-5L questionnaire is a self assessed quality of life questionnaire. The scale measures quality of life on a 5 component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The rater selects a number between 1-100 to describe the condition of their health, 100 being the best imaginable.
Behavioral: PROMIS Cognitive Function 4a Questionnaire — The PROMIS measures function, symptoms, behavior and feelings.
Behavioral: Comprehensive Score for Financial Toxicity (COST) measure — The COST is a questionnaire made up of 11 statements around topics including costs, concerns and resources and is designed to measure financial toxicity. The user answers questions about their concern over finances numbered from 0-4, with 0 being not at all and 4 being very much.

SUMMARY:
The purpose of the study is to assess self-reported side effects and neurocognitive (brain, mood and thinking) functioning among patients treated with commercial axi-cel therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diffuse large b-cell lymphoma, primary mediastinal b-cell lymphoma or transformed follicular lymphoma
* Scheduled to receive commercial axi-cel at Moffitt Cancer Center
* Able to speak and read standard english
* Have no documented or observable psychiatric or neurological diagnoses that interfere with study participation (e.g., schizophrenia)
* Have no history of traumatic brain injury, stroke, or dementia
* Able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to receive axi-cel therapy at Moffitt Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in total neuropsychological performance after axi-cel therapy - Memory | Prior to therapy, then at 30, 90 and 360 days
  Memory changes will be assessed with the Repeatable Battery for the Assessment of Status (RBANS) which assesses immediate memory (list learning and story memory), visuospatial/constructional abilities (figure copy and line orientation), language (picture naming and semantic fluency), attention (digit span and coding), and delayed memory (list recall, list recognition, story recall, and figure recall) domains. Both total scores and scaled/percentile group scores are calculated for each test and total scores are derived for each cognitive domain. Total scores for each cognitive domain are then summed together to create a total scale score.
Change in total neuropsychological performance after axi-cel therapy - Attention and Concentration | Prior to therapy, then at 30, 90 and 360 days
  Attention and concentration are will be assessed using Part 1 of the Color Trails Test (CTT-1) and the Connors Continuous Performance Test Third Edition (CPT3). The CTT is an analogue of the original Trail Making Test without significant influence of language. CTT-1 consists of a page with scattered circles numbered from 1 to 25.
  Even numbered circles are colored yellow and odd-numbered ones are colored pink.
  Respondents are instructed to connect the circles in consecutive numeric order with a continuous line as quickly as possible. The alternating colors are not mentioned in the instructions. A total score is determined by recording the number of seconds required to complete the task.
Change in total neuropsychological performance after axi-cel therapy - Executive Functioning | Prior to therapy, then at 30, 90 and 360 days
  Executive Functioning will be assessed using Part 2 of the Color Trails Test (CTT-2) and the Stroop Color and Word Test. The CTT-2 consists of a page containing 25 pink circles and 25 yellow circles numbered 1 - 50. Participants connect the circles in consecutive order while alternating colors (1 pink, 2 yellow, 3 pink, etc.). A total score is determined by recording the number of seconds required to complete the task. The Stroop Color and Word Test consists of three tasks, a Word Task, a Color Task, and a Color-Word Task. In the Word Task, participants are required to read a list of color words printed in black ink. In the Color Task, participants are presented with rows of X's printed in colored ink, and asked to name the color of each set of X's. In the Color-Word Task, color names are presented in different color ink, and participants are asked to identify the color ink in which each color name is printed. The Stroop yields a score on each task as well as an interference score.
Change in total neuropsychological performance after axi-cel therapy - Hand grip strength | Prior to therapy, then at 30, 90 and 360 days
  The hand grip test assesses hand and forearm strength using a hand dynamometer. Participants without a history of arthritis or hand surgery will be asked to squeeze the dynamometer twice using each hand for a total of two bilateral measurements.
Change in patient-reported outcomes after axi-cel therapy -PROMIS-29 Questionnaire | Prior to therapy, then at 30, 90 and 360 days
  Change in patient-reported outcomes measured using the Patient Reported Outcomes Measurement Information System-29 (PROMIS-29) Questionnaire, which is a 29 item questionnaire assessing aspects of quality of life in the past 7 days on 7 4-item subscales: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance and ability to participate in social activities. Patients rate functioning on a 5-point Likert scale. Higher scores indicate more of the attribute being measured.
Change in patient-reported outcomes after axi-cel therapy - EORTC-QOL Questionnaire | Prior to therapy, then at 14, 30, 60, 90 180 and 360 days
  Change in patient-reported outcomes measured using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) which assess quality of life and symptomatology in the past week using a 4 point Likert scale (1=not at all, 4=very much). Higher scores on the quality of life subscales indicate better quality of life. Higher scores on the symptom items and subscales indicate greater symptomatology.
Change in patient-reported outcomes after axi-cel therapy - QOL Questionnaire | Prior to therapy, then at 7, 14, 30, 60, 90, 180 and 360 days
  Change in patient-reported outcomes measured using the Quality of Life (EQ-5D-5L) Questionnaire, which is a 5-item measure that can be used to describe and value current overall health consisting of 5 items assessing mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Participant chooses from 1 of 5 categories (e.g.; "I have no problems washing or dressing myself" to "I am unable to wash or dress myself"). Higher scores indicate worse overall health.
Change in patient-reported outcomes after axi-cel therapy - Everyday Cognition Questionnaire | Prior to therapy, then at 30, 90 and 360 days
  Change in patient-reported outcomes measured using the Everyday Cognition Questionnaire (ECog) assess the subjective evaluation of cognitive function in routine daily activities. 40 items yield scores for 7 domains (Everyday Memory, Language, Visuospatial Abilities, Planning, Organization, and Divided Attention) and a total score. Items evaluate current cognition compared to 10 years ago; responses are evaluated on a 5-point Likert scale ("better or no change" to "consistently much worse") Higher scores indicate worse subjective cognitive function.
Change in patient-reported outcomes after axi-cel therapy - PROMIS 4a Questionnaire | Prior to therapy, then at 30, 90 and 360 days
  Change in patient-reported outcomes measured using the PROMIS Cognitive Function 4a Questionnaire asks about cognition in the past 7 days using a 5-point Likert scale (1=very often, several times a day; 5=never). Higher scores indicate better overall perceived cognition.
Change in patient-reported outcomes after axi-cel therapy - Comprehensive Score for Financial Toxicity | Prior to therapy, then at 90 days
  Change in patient-reported outcomes measured using the Comprehensive Score for Financial Toxicity (COST). Financial toxicity is assessed using an 11-item patient-reported measure of financial stress used in cancer patients. The COST yields a total score with higher scores indicating less financial toxicity in the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Jim, PhD, Principal Investigator — Moffitt Cancer Center; Fred Locke, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided